CLINICAL TRIAL: NCT04454437
Title: A Phase IIb, Single Arm, Multicenter Trial of Sacituzumab Govitecan in Chinese Patients With Metastatic Triple-negative Breast Cancer Who Received at Least Two Prior Treatments
Brief Title: Study of Sacituzumab Govitecan in Chinese Patients With Metastatic Triple-negative Breast Cancer Who Received at Least Two Prior Treatments
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVER-132-001; CTR20200914 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform)
Record Dates: First submitted 2020-06-05; First posted 2020-07-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan-hziy (Experimental): Participants will receive sacituzumab govitecan-hziy 10 mg/kg on Days 1 and 8 of a 21-day cycle. Participants will continue treatment until disease progression or intolerable toxicity or consent withdrawal for any reason.
  Interventions: Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132

SUMMARY:
The goal of this study is to learn more about the effectiveness of the study drug, sacituzumab govitecan-hziy, in Chinese participants with metastatic triple-negative breast cancer (mTNBC) who received at least 2 systemic chemotherapy regimens.

DETAILED DESCRIPTION:
This is a Phase IIb, single arm, multicenter study of sacituzumab govitecan-hziy in locally advanced or metastatic TNBC patients who are refractory or relapsing after at least 2 prior standard chemotherapy regimens for unresectable, locally advanced or metastatic breast cancer, and these regimens will qualify regardless of triple-negative status at the time they were given. The primary endpoint of the trial will be the objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1) by Independent Review Committee (IRC) in all treated patients.

Participants will be treated until progression requiring discontinuation of further treatment, unacceptable toxicity, study withdrawal, or death, whichever comes first. Tumor response and progression will be assessed using RECIST v 1.1 and assessment by Investigator at the trial center will be sufficient for decisions on continuation of treatment. An independent analysis of response will also be performed by IRC, but this will not be used to make treatment decisions. All participants will visit the Investigator at regular intervals for assessment of safety parameters and adverse events.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female Chinese, 18 years of age or older providing written informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Histologically or cytologically confirmed Triple-negative Breast Cancer (TNBC).
4. Refractory to or relapsed after at least 2 prior standard of care chemotherapy regimens for unresectable, locally advanced or metastatic breast cancer.
5. Measurable disease by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
6. Availability of archival tumor tissue or newly acquired biopsy (FFPE block or a minimum of number 10 unstaining tumor slides, recommended from recurrent or metastatic sites).
7. For individuals with a documented germ-line BRCA1/BRCA2 mutation who received an approved PARP inhibitor, the PARP inhibitor can be used to meet the criteria for one of 2 prior standard of care chemotherapies.
8. All individuals must have been previously treated with a taxane regardless of disease stage (adjuvant, neoadjuvant or advanced) when it was given. Individuals who have contraindications or are intolerant to taxanes are eligible provided that they received at least 1 cycle of a taxane and showed contraindications or intolerance during or at the end of that cycle.
9. Adequate bone marrow, hepatic and renal function, defined as:

   * hemoglobin > 9 g/dL, absolute neutrophil count > 1,500 per mm^3, platelets > 100,000 per mm^3.
   * creatinine clearance of > 60 ml/min calculated using Cockcroft-Gault equation.
   * bilirubin ≤ 1.5 Upper Limit of Normal (ULN), aspartate amino transferase and alanine amino transferase ≤ 2.5 × ULN or ≤ 5 × ULN if known liver metastases and serum albumin ≥ 3 g/dL.
10. Recovered from all prior treatment-related toxicities to Grade 1 or less by National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0) (except alopecia or peripheral neuropathy that may be Grade 2 or less).
11. Individuals must have completed all prior cancer treatments at least 2 weeks prior to the first dose including chemotherapy (includes also endocrine treatment), radiotherapy and major surgery. Prior antibody treatment for cancer must have been completed at least 3 weeks prior to the first dose.
12. Individuals must have at least a 3-month life expectancy.

Key Exclusion Criteria:

1. Previous treatment with topoisomerase 1 inhibitors as a free form or as other formulations.
2. Individuals with a history of or current central nervous system (CNS) metastases. A scan to confirm the absence of brain metastases is not required. Individuals with unknown CNS metastatic status and any clinical signs indicative of CNS metastases are eligible if CNS metastases are excluded using CT and/or MRI scans.
3. Individuals with Gilbert's disease.
4. Individuals with non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while individuals with other prior malignancies must have had at least a 3-year disease-free interval.
5. Individuals known to be human immunodeficiency virus positive.
6. Individuals with active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. In individuals with a history of HBV, hepatitis B core antibody (HBcAb) testing is required and if positive, then HBV DNA testing will be performed and if positive the individual will be excluded.
7. Known history of unstable angina, myocardial infarction (MI), or chronic heart failure present within 6 months of first dose or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy or left ventricular ejection fraction < 50%.
8. Known history of clinically significant active chronic obstructive pulmonary disease, or other moderate-to-severe chronic respiratory illness present within 6 months of the first dose.
9. Infection requiring systematic antibiotic use within 1 week of the first dose.
10. Individuals with active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease) and individuals with a history of bowel obstruction or gastrointestinal (GI) perforation.
11. High dose systemic corticosteroids within 2 weeks prior to the first dose (however, low dose corticosteroids ≤ 10 mg prednisone or equivalent daily are permitted provided the dose is stable for 4 weeks).
12. Scheduled surgery during the study, other than minor surgery which would not delay study treatment.
13. Individuals who have received a live vaccine within 30 days of first dose.
14. Rapid deterioration during Screening prior to the first dose, eg, significant change in performance status, unstable pain symptoms requiring modifications in analgesic management.
15. Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
16. Females who are pregnant or lactating.
17. Females of childbearing potential or fertile males unwilling to use highly effective* contraception during study and up to 6 months after treatment discontinuation in females of childbearing potential and 3 months in males post last Investigational Medicinal Product (IMP) administration.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1) By Independent Review Committee (IRC) | Up to 3 years
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) by IRC | Up to 3 years
  DOR is defined as the time between the date until the earlier date of disease progression or death.
Clinical Benefit Rate (CBR) | Up to 3 years
  CBR is defined as best overall response of CR or PR or stable disease (SD) of at least 6 months.
Progression-free Survival (PFS) | Up to 3 years
  PFS is defined as the time since the first dose of trial treatment until the earlier date of disease progression as defined by RECIST v1.1 or death due to any cause.
Overall survival (OS) | Up to 3 years
  OS is defined as the time since the first dose of trial treatment until death due to any cause.
Percentage of Participants Experiencing Adverse Events (AEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | First dose date up to 3 years plus 30 days
Percentage of Participants Experiencing Serious Adverse Events (SAEs) According to NCI CTCAE Version 5.0 | First dose date up to 3 years plus 30 days
Pharmacokinetic (PK) Parameter: Cmax of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 3 years
  Cmax is defined as the maximum observed concentration of drug.
Percentage of Participants Who Developed Anti-Drug Antibodies (ADAs) Against Sacituzumab Govitecan-hziy | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (17):
- China (17):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Chinese PLA General Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Sun Yat-sen University, Cancer Center, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu B, Ma F, Wang T, Wang S, Tong Z, Li W, Wu X, Wang X, Sun T, Pan Y, Yao H, Wang X, Luo T, Yang J, Zeng X, Zhao W, Cong XJ, Chen J. A Phase IIb, single arm, multicenter trial of sacituzumab govitecan in Chinese patients with metastatic triple-negative breast cancer who received at least two prior treatments. Int J Cancer. 2023 May 15;152(10):2134-2144. doi: 10.1002/ijc.34424. Epub 2023 Jan 30. PMID 36621000
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT04454437